CLINICAL TRIAL: NCT01232556
Title: AN OPEN-LABEL, RANDOMIZED, PHASE 3 STUDY OF INOTUZUMAB OZOGAMICIN ADMINISTERED IN COMBINATION WITH RITUXIMAB COMPARED TO DEFINED INVESTIGATOR'S CHOICE THERAPY IN SUBJECTS WITH RELAPSED OR REFRACTORY CD22-POSITIVE AGGRESSIVE NON-HODGKIN LYMPHOMA WHO ARE NOT CANDIDATES FOR INTENSIVE HIGH-DOSE CHEMOTHERAPY
Brief Title: A Study Of Inotuzumab Ozogamicin Plus Rituximab For Relapsed/Refractory Aggressive Non-Hodgkin Lymphoma Patients Who Are Not Candidates For Intensive High-Dose Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely on May 16, 2013, for futility. No new or unexpected safety issues were identified.
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1931008; 3129K5-3303 (Other: Alias Study Number); 2010-020147-12 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-11-02 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: inotuzumab ozogamicin; aggressive Non-Hodgkin lymphoma; diffuse large b-cell lymphoma; relapsed/refractory lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Inotuzumab Ozogamicin; Rituximab; Gemcitabine

ARMS (2):
- 1 (Experimental): Inotuzumab ozogamicin+rituximab
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Rituximab
- 2 (Active Comparator): Investigator's choice of (1) rituximab+gemcitabine, or (2) rituximab+bendamustine
  Interventions: Drug: rituximab + gemcitabine; Drug: rituximab +bendamustine

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — 1.8 mg/m2 on day 2 every 28 days by IV infusion, 3 to 6 cycles
  Other Names: CMC-544
  Arms: 1
Drug: Rituximab — 375 mg/m2 on day 1 every 28 days by IV infusion, 3 to 6 cycles
  Arms: 1
Drug: rituximab + gemcitabine — rituximab 375 mg/m2 on days 1, 8, 15, and 22 of cycle 1, and day 1 of cycles 2 to 6, every 28 days by IV infusion, 3 to 6 cycles; gemcitabine 1000 mg/m2 on days 1, 8, and 15 every 28 days, 3 to 6 cycles
  Arms: 2
Drug: rituximab +bendamustine — rituximab 375 mg/m2 on day 1 every 28 days by IV infusion, 3 to 6 cycles; bendamustine 120 mg/m2 on days 1 and 2 by IV infusion every 28 days, 3 to 6 cycles
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of inotuzumab ozogamicin plus rituximab in relapsed/refractory aggressive Non-Hodgkin lymphoma patients who are not candidates for intensive high-dose chemotherapy. Specifically, the goal is to demonstrate the superiority of this combination compared with an active comparator arm (investigator's choice of rituximab+bendamustine or rituximab+gemcitabine) using the primary endpoint of overall survival.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2014-03-28 (Actual); Study Completion 2014-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (174):
- United States (79):
  - Disney Family Cancer Center at Providence St Joseph Medical Center, Burbank, California
  - Providence St Joseph Medical Center, Burbank, California
  - Hematology-Oncology Medical Group of Fresno Inc, Fresno, California
  - Ronald Reagan UCLA Medical Center Drug Information Center Department of Pharmaceutical Services, Los Angeles, California
  - Clinical Research Unit, Los Angeles, California
  - Peter Morton Medical Plaza, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Sansum Clinic, Santa Barbara, California
  - UCLA Santa Monica Hematology Oncology, Santa Monica, California
  - Sansum Clinic, Solvang, California
  - Howard University Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - 21st Century Oncology of Jacksonville, LLC, Fernandina Beach, Florida
  - Davis Cancer Pavilion and Shands Medical Plaza, Gainesville, Florida
  - Shands Cancer Hospital at the University of Florida, Gainesville, Florida
  - UF Health Davis Cancer Pavillion and Shands Med Plaza, Gainesville, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - 21st Century Oncology of Jacksonville, LLC, Jacksonville, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - 21st Century Oncology of Jacksonville, Inc., Jacksonville, Florida
  - Medical Specialists Of The Palm Beaches, Lake Worth, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Mercy Hospital, Miami, Florida
  - Mercy Research Institute, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology of Jacksonville, LLC, Orange Park, Florida
  - Georgia Regents Medical Cancer Pharmacy, Augusta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Decatur Memorial Hospital (DMH), Decatur, Illinois
  - Floyd Memorial Cancer Center of Indiana, New Albany, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - University of Kentucky A.B. Chandler Medical Center, Lexington, Kentucky
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute at farmington Hills, Farmington Hills, Michigan
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Barnes-Jewish St. Peters, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University in St Louis, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, P.C. d/b/a Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Beth Israel Medical Center;, New York, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - St Luke's- Roosevelt Hospital Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, The Cancer Center, Stony Brook, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University Hospital, Cincinnati, Ohio
  - West Chester Hospital Medical Building, West Chester, Ohio
  - OU Medical Center Presbyterian Professional Building, Oklahoma City, Oklahoma
  - OU Medical Center Presbyterian Tower, Oklahoma City, Oklahoma
  - Peggy and Charles Stephenson Cancer Center (chemo & infusion), Oklahoma City, Oklahoma
  - Peggy and Charles Stephenson Cancer Center (clinic location), Oklahoma City, Oklahoma
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - Good Samaritan Hospital, Corvallis, Corvallis, Oregon
  - Samaritan Ambulatory Infusion Services, Corvallis, Oregon
  - Samaritan Pacific Coast Hospital, Newport, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Guthrie Clinic, Ltd., Sayre, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Thompson Oncology Group, Knoxville, Tennessee
  - Thompson Oncology Group, Maryville, Tennessee
  - Thompson Oncology Group, Sevierville, Tennessee
  - University Hospital - St. Paul, Dallas, Texas
  - University Hospital - Zale Lipshy, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor: Charles A. Sammons Cancer Center, Dallas, Texas
  - Simmons Comprehensive Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (6):
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams Brabant
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
  - St Augustinus Ziekenhuis, Wilrijk
  - Cliniques universitaires UCL de Mont-Godinne,, Yvoir
- Bulgaria (3):
  - UMBAL Sveti Georgi, Klinika po hematologia, Plovdiv
  - SBAL na Hematologichnichni Zabolyavania,CTH Sofia, Sofia
  - Spetsializirana Bolnitsa za Aktivno Lechenie na Hematologichni Zabolyavania, CTH Sofia, Sofia
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Hopital Fleurimont, Sherbrooke, Quebec
- Croatia (2):
  - University Hospital Zagreb, Zagreb
  - University Hospital Dubrava Department of Internal Medicine Division of Hematology, Zagreb
- Czechia (2):
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Czech Republic
  - Fakultni nemocnice Brno, Brno
- France (8):
  - Département Pharmacie, Marseille, Bouches-du-rhône
  - Institut Paoli Calmettes, Marseille, Cedex 09
  - Hopital Andre Mignot, Le Chesnay, Yvelines
  - Hospital Universitaire Andre Mignot, Le Chesnay, Yvelines
  - Centre Leon Berard, Lyon
  - CHU Saint Eloi, Montpellier
  - Hopital du haut Leveque, Pessac
  - Centre Henri Becquerel, Rouen
- Germany (7):
  - Universitaetsklinikum Aachen, Aachen
  - Sozialstiftung Bamberg, Bamberg
  - Charite Campus Benjamin Franklin, Berlin
  - Charite Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Mainz, Mainz
  - TU Muenchen III. Medizinische Klinik, München
  - Universitaetsklinik Ulm, Ulm
- Hungary (3):
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz /, Budapest
  - DEOEC, Belgyogyaszati Intezet, Debrechen
  - Somongy Megyei Kaposi Mor Okato Korhaz/ Belgyogyaszati osztaly, Kaposvár
- India (4):
  - Kodlikeri Memorial Hospital, Aurangabad, Maharashtra
  - Sahyadri Clinical Research and Development Center, Pune, Maharashtra
  - OEC Record Management Company Pvt. Ltd.,, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
- Bon Secours Hospital, Cork, Ireland
- Japan (13):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Gunma University Hospital, Maebashi, Gunma
  - Tohoku University Hospital, Sendai, Miyagi
  - Matsushita Memorial Hospital, Moriguchi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
  - Akita University Hospital, Akita
  - National Kyushu Cancer Center, Fukuoka
  - Tokai University Hospital, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
- Klaipeda Seamen's Hospital, Public Institution, department of Oncology, Klaipėda, Lithuania
- Instituto Biomédico de Investigación A.C., Aguascalientes, Aguascalientes. Mexico, Mexico
- Poland (2):
  - Niepubliczny Zaklad Opieki Zdrowotnej AVI Diagnostyka Obrazowa, Warsaw
  - Klinika Nowotworow Ukladu Chlonnego, Warsaw
- Puerto Rico (2):
  - Advanced Infusion Services, Cataño
  - Hospital Espanol Auxilio Mutuo de Puerto Rico Inc, San Juan
- Russia (3):
  - Federal State Budgetary Institution Hematology Scientific Centre of Ministry of, Moscow
  - Moscow State Healthcare Institution City clinical hospital S.P. Botkin, Moscow
  - Institute of Pediatric Hematology and Transplantology R.M.Gorbacheva, Saint Petersburg
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Narodny onkologicky ustav, Bratislava, Slovakia
- Spain (7):
  - Hospital Virgen Del Rocio, Seville, Andalusia
  - Hospital Universitario De Salamanca, Salamanca, Castille and LION
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Institut Catala d'Oncologia-L'Hospitalet, L'Hospitalet de Llobregat (bcn)
  - Hospital Universitario de Canarias, La Laguna (Tenerife)
  - Hospital de la Princesa, Madrid
- Sweden (2):
  - Universitetssjukhuset, Linköping
  - Skanes Universitetssjukhus i Lund, Lund
- Taiwan (4):
  - Chang Gung Medical Foundation - Linkou Branch, Kuei-Shan Hsiang, Taoyuan County
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Department of Internal Medicine, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (2):
  - Hematology Division Department of Medicine Faculty of Medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok
  - Chiang Mai University, Chiang Mai
- Ukraine (3):
  - Regional Treatment and Diagnostic Hematology Center Communal Establishment, Cherkasy
  - Department of Oncology and Medical Radiology of State Institution, Dnipropetrovsk
  - SI"Research Center for Radiation Medicine of NAMS of Ukraine", Kyiv
- United Kingdom (12):
  - Barts Cancer Centre Dept Haemato-oncology St. Bartholomew's Hospital Barts Health NHS Trust, London
  - Chemotherapy Preparative Unit St. Bartholomew's Hospital, London
  - Department of Medical Oncology St. Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester
  - Department of Clinical Pathology Newcastle upon Tyne Hospitals NHS Foundation Trust Royal Victoria I, Newcastle upon Tyne
  - Department of Clinical Biochemistry Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - Northern Centre for Cancer Care, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - Pathology Department Nottingham University Hospital - City Hospital Campus, Nottingham
  - Pharmacy Nottingham University Hospital - City Hospital Campus, Nottingham
  - Local Laboratory Nottingham University Hospital - City Hospital Campus, Nottingham
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1931008&StudyName=%20A%20Study%20Of%20Inotuzumab%20Ozogamicin%20Plus%20Rituximab%20For%20Relapsed/Refractory%20Aggressive%20Non-Hodgkin%20Lymphoma%20Patients%20Who%20Are%20Not%20Candidates%20F

RESULTS

PARTICIPANT FLOW:
Groups:
- Inotuzumab Ozogamicin Plus (+) Rituximab: Participants received rituximab 375 milligrams per square meter (mg/m^2) via intravenous (IV) infusion on Day 1 and inotuzumab ozogamicin 1.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for a maximum of 6 cycles.
- Rituximab+Gemcitabine or Rituximab+Bendamustine: Participants received either R-bendamustine (rituximab 375 mg/m^2 via IV infusion on Day 1 and bendamustine 120 mg/m^2 via IV infusion on Days 1 and 2 in 28-day cycles for a maximum of 6 cycles) or R-gemcitabine (rituximab 375 mg/m^2 via IV infusion on Days 1, 8, 15 and 22 of Cycle 1 and on Day 1 for all other cycles, and gemcitabine 1000 mg/m^2 via IV infusion on Days 1, 8 and 15 of each 28-day cycle for a maximum of 6 cycles). Choice of therapy was at the discretion of the investigator.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin Plus (+) Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Started | 166 | 172
Treated | 165 (One subject in this arm received rituximab only and was excluded from the safety population.) | 167
Completed | 7 | 1
Not Completed | 159 | 171
Not completed — Withdrawal by Subject | 21 | 17
Not completed — Death | 97 | 97
Not completed — Lost to Follow-up | 0 | 2
Not completed — Terminated by Sponsor | 35 | 51
Not completed — Other | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population - included all participants who are randomized into the study.
Groups:
- Inotuzumab Ozogamicin+Rituximab: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for a maximum of 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine | Total
Number analyzed (Participants) | 166 | 172 | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age measure using mean with Standard deviation
  Years | 68.6 (12.29) | 66.9 (11.40) | 67.7 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 75 | 75 | 150
    Male | 91 | 97 | 188

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause, censoring at the date of last contact or the end of the study. The Kaplan-Meier method was used to determine OS. The hazard ratio and corresponding 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: From randomization up to 5 years after last dose or up to final study visit, whichever occurs first.
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Months | 9.5 [7.0 to 14.5] | 9.5 [7.7 to 14.1]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Primary null hypothesis: Equality of survival distributions. Sample size sufficient to have power 0.96 for an experimental/control hazard ratio of 0.6; Test type: Superiority or Other; p = 0.708, Log Rank — A one sided 0.025 level testing plan was specified with two interim analyses and final testing level at one-sided 0.023; From one sided stratified log-rank test; Hazard Ratio (HR) = 1.083, 95% CI 2-sided [0.82 to 1.44] — From stratified Cox proportional hazards model. The stratification factors are are pre-randomization investigator choice, baseline Secondary International Prognostic Index (sIPI), and best response to most recent chemo therapy

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from date of randomization to date of progressive disease (PD, including investigator's claim of clinical progression), date of death from any cause, or initiation of a new treatment for the lymphoma due to persistent/refractory disease. The Kaplan-Meier method was used to determine PFS. The hazard ratio and corresponding 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
  PD requires the following:
  1. Appearance of any new lesion more than 1.5 cm in any axis during or at the end of treatment, even if other lesions are decreasing in size.
  2. At least a 50% increase from nadir in the sum of the product diameters of any previously involved nodes, or in a single involved node, or the size of other lesions.
  3. At least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis.
Time Frame: From randomization up to 2 years or final study visit, whichever occurs first, including but not limited to planned assessments scheduled approximately every 12 weeks.
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Months | 3.7 [2.9 to 5.0] | 3.5 [2.8 to 4.9]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Second comparison in hierarchical testing strategy was used for power calculation; Test type: Superiority or Other; p = 0.271, Log Rank — An hierarchical testing strategy was specified for OS, PFS and response. PFS could be tested at the 0.023 level if the OS test result were positive. Response could be tested if both the OS and PFS test results were positive; From one sided stratified log-rank test; Hazard Ratio (HR) = 0.924, 95% CI 2-sided [0.72 to 1.19] — From stratified Cox proportional hazards model. The stratification factors are are pre-randomization investigator choice, baseline sIPI, and best response to most recent chemo therapy

3. Secondary Outcome: Percentage of Participants With A Best Overall Response of CR or Partial Response (PR) Per NCI International Response Criteria for NHL
Description: CR is defined as disappearance of all detectable clinical evidence of disease (including cleared infiltrate on repeat bone marrow aspirate/biopsy if lymphoma involvement of bone marrow before treatment).
  Partial Response (PR) requires the following:
  1. ≥50 % decrease in SPD of the six largest dominant nodes or nodal masses.
  2. No increase in the size of other nodes, liver, or spleen.
  3. Splenic and hepatic nodules must regress by ≥50% in the SPD, or for single nodules, in the greatest transverse diameter.
  4. With the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present.
  5. No new sites of disease. The 95% CI was determined using the exact method based on binomial distribution.
Time Frame: Up to 2 years from first study drug dose or up to final study visit, whichever occurs first, including but not limited to planned assessments scheduled approximately every 12 weeks.
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Percentage of Participants | 29.5 [22.70 to 37.08] | 29.7 [22.94 to 37.08]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Third comparison in hierarchical testing strategy was used for power calculation; Test type: Superiority or Other; p = 0.843, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; The stratification factors are pre-randomization investigator choice, baseline sIPI, and best response to most recent chemo therapy

4. Secondary Outcome: Percentage of Participants With A Best Overall Response of CR, Unconfirmed CR (unCR), PR, or Unconfirmed PR (unPR) Per NCI International Response Criteria for NHL
Description: CR is defined as disappearance of all detectable clinical evidence of disease (including cleared infiltrate on repeat bone marrow aspirate/biopsy if lymphoma involvement of bone marrow before treatment).
  Partial Response (PR) requires the following:
  1. ≥50 % decrease in SPD of the six largest dominant nodes or nodal masses.
  2. No increase in the size of other nodes, liver, or spleen.
  3. Splenic and hepatic nodules must regress by ≥50% in the SPD, or for single nodules, in the greatest transverse diameter.
  4. With the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present.
  5. No new sites of disease. unCR and unPR means didn't have confirmatory assessment (including bone marrow assessment for CR).
  The 95% CI was determined using the exact method based on binomial distribution.
Time Frame: as for outcome 3
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Percentage of Participants | 41.0 [33.40 to 48.85] | 43.6 [36.07 to 51.36]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Third comparison in hierarchical testing strategy was used for power calculation; Test type: Superiority or Other; p = 0.714, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the first date of response until the first date that the progressive disease (PD) or death is objectively documented. The hazard ratio and corresponding 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: as for outcome 3
Population: ITT population; only participants with a CR, unCR, PR, or unPR were included in the analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Months | 11.56 [7.8 to NA] — The upper limit of the 95 percent (%) confidence interval could not be determined due to the large number of censored events. | 6.93 [5.5 to 10.8]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; DOR was not part of the formal hypothesis testing strategy; Test type: Superiority or Other; p = 0.142, Log Rank; From one sided stratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.47 to 1.25] — From stratified Cox proportional hazards model. The stratification factors are pre-randomization investigator choice, baseline sIPI, and best response to most recent chemo therapy

6. Secondary Outcome: Health Status as Assessed by the European Quality of Life 5 Dimension (EQ-5D) Questionnaire
Description: EQ-5D consists of a descriptive system and an EQ visual analogue scale. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The scale, the best state is marked 100 and the worst state is marked 0, is to help the participant to say how good or bad a health state is. EQ-5D index, which was reported, was derived based on US weight. The range of EQ-5D index is -0.109 to 1.00. Higher scores mean better outcomes. The average post-baseline scores for EQ-5D index were computed at approximately Week 12. The overall treatment comparisons were estimated at approximately Week 12.
Time Frame: Assessed at Day 1 of each cycle and 6-9 weeks after the last dose, Cycle 3 (Week 12) reported
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Unit on a scale | 0.79 [0.76 to 0.82] | 0.77 [0.74 to 0.79]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Test type: Superiority or Other; p = 0.2892, Mixed Models Analysis; Repeated measures mixed effects model with treatment, time, treatment-by-time interaction, and baseline as covariate; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.06]

7. Secondary Outcome: Health Related Quality of Life as Assessed by the Functional Assessment of Cancer Therapy for Lymphoma (FACT-Lym) Questionnaire
Description: FACT-Lym is a questionnaire that begins with 27 items covering four core Health-Related Quality of Life subscales: Physical Well-being (7 items), Social/Family Well-being (7), Emotional Well-being (6), and Functional Well-being (7). The FACT-Lym also includes an additional concerns subscale (15 items). It also asks participants about their concerns about lumps and swelling, fevers, infections, weight, appetite, emotional stability and treatment. The participants were requested to circle one number on a 0 to 4 points scale per line to indicate how true each statement has been for him/her during the past 7 days. FACT-Lym total score, which was reported, was derived based on FACT-Lym scoring guideline (Version 4). The range of FACT-Lym total score is 0 to 168. Higher scores mean better outcomes. The average post-baseline FACT-Lym total scores were computed at approximately Week 12. The overall treatment comparisons were estimated at approximately Week 12.
Time Frame: Assessed at Day 1 of each cycle and 6-9 weeks after the last dose, Cycle 3 (Week 12) reported
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 166 | 172
Unit on a scale | 120.07 [116.74 to 123.41] | 116.96 [113.74 to 120.19]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin+Rituximab vs Rituximab+Gemcitabine or Rituximab+Bendamustine; Test type: Superiority or Other; p = 0.1879, Mixed Models Analysis; Repeated measures mixed effects model with treatment, time, treatment-by-time interaction, and baseline as covariate; Mean Difference (Final Values) = 3.11, 95% CI 2-sided [-1.52 to 7.74]

8. Primary Outcome: Percentage of Participants With a Treatment Emergent Adverse Event (TEAE) (Safety Population)
Description: Includes all TEAEs: Any event that occurred after the first dose of study drug and was not present prior to study drug administration or worsened in severity after study drug administration..
Time Frame: Up to 20 weeks after the first dose of study drug
Population: Safety Population - included all participants who received at least 1 dose of test article (either inotuzumab ozogamicin administrated in combination with rituximab or investigator's choice). This population only excluded participants who never received any test article.
Measure: Number; unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Number analyzed (Participants) | 164 | 167
Percentage of Participants
  % participants with a TEAE | 98.8 | 100.0
  % participants with serious TEAE | 37.2 | 37.7
  % participants with Grade 3 or 4 TEAE | 79.9 | 79.6
  % participants with Grade 5 TEAE | 14.6 | 13.8
  % participants for study drug discontinuation | 25.0 | 18.0
  % participants with dose reductions due to TEAEs | 27.4 | 29.3
  % participants for study drug stopped temporarily | 31.1 | 46.1

ADVERSE EVENTS:
Time Frame: Up to 22 weeks after the informed consent
Description: Adverse Events calculated using safety population. One subject in the rituximab+ inotuzumab ozogamicin arm received rituximab only, and was excluded from the safety population analysis. AE summaries below are inclusive of AEs from first dose date up to 56 days after last dose of study drug.
Arm/Group | Inotuzumab Ozogamicin+Rituximab | Rituximab+Gemcitabine or Rituximab+Bendamustine
Serious Adverse Events (participants affected / at risk) | 61/164 | 63/167
Other Adverse Events (participants affected / at risk) | 155/164 | 158/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin+Rituximab (N=164) | Rituximab+Gemcitabine or Rituximab+Bendamustine (N=167)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 2
Disease progression (General disorders) | 15 | 20
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 0
Oedema due to hepatic disease (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 4
Sudden death (General disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium febrile (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin+Rituximab (N=164) | Rituximab+Gemcitabine or Rituximab+Bendamustine (N=167)
Anaemia (Blood and lymphatic system disorders) | 24 | 43
Leukopenia (Blood and lymphatic system disorders) | 37 | 54
Lymphopenia (Blood and lymphatic system disorders) | 28 | 39
Neutropenia (Blood and lymphatic system disorders) | 57 | 81
Thrombocytopenia (Blood and lymphatic system disorders) | 101 | 64
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 10
Abdominal pain (Gastrointestinal disorders) | 14 | 13
Constipation (Gastrointestinal disorders) | 38 | 33
Diarrhoea (Gastrointestinal disorders) | 22 | 31
Nausea (Gastrointestinal disorders) | 50 | 54
Vomiting (Gastrointestinal disorders) | 23 | 32
Asthenia (General disorders) | 13 | 14
Chills (General disorders) | 5 | 9
Fatigue (General disorders) | 55 | 42
Oedema peripheral (General disorders) | 17 | 15
Pyrexia (General disorders) | 37 | 35
Nasopharyngitis (Infections and infestations) | 9 | 6
Urinary tract infection (Infections and infestations) | 9 | 12
Alanine aminotransferase increased (Investigations) | 28 | 17
Aspartate aminotransferase increased (Investigations) | 44 | 18
Blood alkaline phosphatase increased (Investigations) | 24 | 16
Blood bilirubin increased (Investigations) | 10 | 4
Blood creatinine increased (Investigations) | 5 | 13
Blood lactate dehydrogenase increased (Investigations) | 9 | 4
Gamma-glutamyltransferase increased (Investigations) | 38 | 16
Haemoglobin decreased (Investigations) | 4 | 10
Platelet count decreased (Investigations) | 9 | 7
Weight decreased (Investigations) | 4 | 11
White blood cell count decreased (Investigations) | 4 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 12 | 3
Decreased appetite (Metabolism and nutrition disorders) | 28 | 31
Hypercalcaemia (Metabolism and nutrition disorders) | 9 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 12
Dizziness (Nervous system disorders) | 8 | 13
Dysgeusia (Nervous system disorders) | 10 | 8
Headache (Nervous system disorders) | 8 | 11
Insomnia (Psychiatric disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Rash (Skin and subcutaneous tissue disorders) | 8 | 13

LIMITATIONS AND CAVEATS:
Interpretation of the results is limited by the small number of subjects analyzed and follow-up period was shortened due to the early termination of the study.

Adverse Events were calculated using the safety populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No